CLINICAL TRIAL: NCT00727571
Title: Prospective Observational Study to Evaluate Physical Performance and Quality of Life in Older Long Stay Nursing Home Residents With Chronic Kidney Disease With and Without Anemia
Brief Title: LEARN-6™: A Prospective, Observational Nursing Home Study
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20050239
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: Anemia; Chronic Kidney Disease; Quality of Life; CKD; Chronic Renal Insufficiency
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — N/A (None Retained)

GROUPS / COHORTS (4):
- No CKD or Anemia: Chronic kidney disease (CKD) is based on estimated Glomerular Filtration Rate (GFR), calculated by the Modification of Diet in Renal Disease (MDRD) method, of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per World Health Organization (WHO) criteria. Participants completed the study after Week 1; data contributed to prevalence estimates.
  Interventions: Other: Observations
- No CKD, but Anemia: CKD is based on estimated GFR calculated by the MDRD method of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per WHO criteria. Participants completed the study at Week 2 and completed an anemia work-up; data contributed to prevalence estimates.
  Interventions: Other: Observations
- CKD with Anemia: CKD is based on estimated GFR calculated by the MDRD method of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per WHO criteria. Participants were observed for 26 weeks and completed an anemia work-up, and mobility and physical performance assessments.
  Interventions: Other: Observations
- CKD with no Anemia: CKD is based on estimated GFR calculated by the MDRD method of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per WHO criteria. Participants were observed for 26 weeks and completed mobility and physical performance assessments.
  Interventions: Other: Observations

INTERVENTIONS:
Other: Observations — This is a non-interventional, observational study; no investigational product is being used

SUMMARY:
This is a prospective, multicenter, observational, hypothesis-generating study exploring mobility, Quality of Life and other physical performance measures among older, long-term stay Nursing Home residents with CKD, with versus without anemia. Enrolled patients will participate in the study up to a total of 26 weeks and be assessed at Weeks 1, 2, 14 and 26/End of Study. Based upon Week 1 hemoglobin and serum creatinine lab results, participants will be categorized into 1 of 4 groups.

DETAILED DESCRIPTION:
Study Design: Multicenter, non-interventional, 26-week, prospective, observational study of older, long-term stay residents with CKD, with and without anemia, in US Nursing Homes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Long-term resident of NH as documented in medical record by Director of Nursing (DON) or Medical Director or as indicated in Minimum Data Set (MDS) Section Q
* Able to walk at least 1 step or propel wheelchair 1 revolution of wheel
* Able to follow a one-step instruction
* Written informed consent

Exclusion Criteria:

* Admitted to NH for short stay rehabilitation (anticipated stay less than 3 months)
* Receiving Renal Replacement Therapy (RRT)
* Major surgery within the past 3 months
* Life expectancy < 6 months or receiving palliative care
* Currently enrolled in or has not yet completed at least 30 days since ending investigational device or drug study(s), or is receiving investigational agent(s)
* Currently is enrolled in an interventional trial
* Previously withdrawn from this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older, long-term stay Nursing Home (NH) residents with CKD, with and without anemia
Sampling Method: Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Binder EF, White HK, Resnick B, McClellan WM, Lei L, Ouslander JG. A prospective study of outcomes of nursing home residents with chronic kidney disease with and without anemia. J Am Geriatr Soc. 2012 May;60(5):877-83. doi: 10.1111/j.1532-5415.2012.03941.x. Epub 2012 May 9. PMID 22568452
- [Background] McClellan WM, Resnick B, Lei L, Bradbury BD, Sciarra A, Kewalramani R, Ouslander JG. Prevalence and severity of chronic kidney disease and anemia in the nursing home population. J Am Med Dir Assoc. 2010 Jan;11(1):33-41. doi: 10.1016/j.jamda.2009.07.003. Epub 2009 Nov 6. PMID 20129213
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 815 patients were enrolled; 21 of these could not be classified into the defined groups because of missing lab values at enrollment. Their anemic/CKD status is therefore not available.
Groups:
- No CKD or Anemia: Chronic kidney disease (CKD) is based on an estimated Glomerular Filtration Rate (GFR), calculated by the Modification of Diet in Renal Disease (MDRD) method, of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per World Health Organization (WHO) criteria. Participants completed the study after Week 1; data contributed to prevalence estimates.
Period: Overall Study
Arm/Group | No CKD or Anemia | CKD With Anemia | CKD With no Anemia | No CKD, But Anemia
Started | 232 | 228 | 165 | 169
Completed | 231 | 173 | 135 | 163
Not Completed | 1 | 55 | 30 | 6
Not completed — Ineligibility determined | 1 | 1 | 1 | 0
Not completed — Death | 0 | 19 | 5 | 1
Not completed — Physician Decision | 0 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 10 | 11 | 0
Not completed — Subject Non Compliance | 0 | 6 | 0 | 4
Not completed — Dismissed from nursing home | 0 | 9 | 5 | 0
Not completed — Hospitalization | 0 | 1 | 0 | 1
Not completed — AE not leading to hospitalization | 0 | 0 | 2 | 0
Not completed — Other | 0 | 4 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- No CKD, But Anemia; CKD With Anemia; CKD With no Anemia: CKD is based on estimated GFR calculated by the MDRD method of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per WHO criteria.
- No CKD or Anemia: CKD is based on estimated GFR, calculated by the MDRD method, of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per WHO criteria.
- Total: Total of all reporting groups
Arm/Group | No CKD, But Anemia | No CKD or Anemia | CKD With Anemia | CKD With no Anemia | Total
Number analyzed (Participants) | 169 | 232 | 228 | 165 | 794
Age, Continuous [Mean (Standard Deviation); unit: Years] | 82.6 (8.3) | 81.6 (8.2) | 84.6 (8.1) | 83.8 (8.4) | 83.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 172 | 159 | 139 | 558
  Male | 81 | 60 | 69 | 26 | 236

OUTCOME MEASURES:

1. Primary Outcome: Total Distance Walked or Wheeled in a Maximum of 10 Minutes at Each Visit
Description: The distance a participant walked, with or without an assistive device and stand-by assistance of 1 person, or propelled him/herself in a wheelchair with or without the use of his/her feet, over level ground, during a period of up to 10 minutes including up to two 30-second rest periods (at weeks 2, 14 and 26).
Time Frame: Weeks 2, 14 and 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Median (Inter-Quartile Range); unit: feet
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 209 | 152
feet
  Week 2 (N=209, 152) | 210.0 [83.4 to 540.0] | 253.1 [91.8 to 540.0]
  Week 14 (N=173, 134) | 210.0 [79.3 to 500.0] | 246.5 [108.0 to 680.0]
  Week 26 (N=158, 124) | 185.0 [87.3 to 450.0] | 198.5 [99.0 to 497.3]

2. Secondary Outcome: Number of Participants With Anemia
Description: Anemia is defined using World Health Organization (WHO) criteria as Hemogloblin <12 g/dL in women, < 13 g/dL in men.
Time Frame: Baseline
Population: All enrolled patients with available anemia lab results.
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 794
participants | 397

3. Secondary Outcome: Percentage of Participants With Anemia Related Conditions at Baseline
Description: The percentages of anemic subjects with iron deficiency, vitamin B12 deficiency, gastrointestinal (GI) bleed, chronic inflammation, and folate deficiency. Anemia of iron deficiency is defined as reduced serum iron, reduced transferrin saturation, ferritin less than 12 ng/mL plus increased Total Iron Binding Capacity (TIBC), per normal laboratory range. Anemia of chronic inflammation defined as reduced serum iron and transferrin saturation, increased or normal ferritin, and reduced or normal TIBC. GI bleed is based on the result of the stool guaiac sample(s) collected: A participant is considered to have GI bleed if one guaiac sample is positive, and not to have GI bleed only if all of his/her three stool guaiac samples were negative.
  Vitamin B12 and folate deficiency based on standard laboratory ranges.
Time Frame: Baseline
Population: Enrolled patients with anemia
Measure: Number; unit: Percentage of participants
Groups:
- No CKD But Anemia: CKD is based on estimated GFR calculated by the MDRD method of < 60 mL/min/1.73m^2. Anemia is defined as Hemogloblin <12 g/dL in women, < 13 g/dL in men per WHO criteria.
Arm/Group | CKD With Anemia | No CKD But Anemia
Number analyzed (Participants) | 228 | 169
Percentage of participants
  Iron deficiency | 0.0 | 0.0
  Vitamin B12 deficiency | 2.6 | 5.3
  Gastrointestinal (GI) Bleed | 11.4 | 10.1
  Chronic inflammation | 21.9 | 18.3
  Folate deficiency | 2.2 | 4.1

4. Secondary Outcome: Estimated Glomerular Filtration Rate (GFR) for Participants With CKD
Description: Estimated GFR measures how much blood the kidneys are filtering, and was calculated using 2 methods: 1. Modification of Diet in Renal Disease study (MDRD) formula: estimated GFR = 186 x [Serum creatinine]^-1.154 x [Age]^-0.203 x [0.742 if patient is female] x [1.210 if patient is black]. 2. Cockcroft-Gault formula: GFR = (140-age) * (Weight in kg) * (0.85 if female) / (72 * Serum Creatinine).
Time Frame: Weeks 1, 14 and 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 228 | 165
mL/min/1.73 m^2
  Week 1 - MDRD (N=228, 165) | 42.1 (10.6) | 44.9 (9.9)
  Week 14 - MDRD (N=183, 143) | 42.6 (11.6) | 48.0 (15.0)
  Week 26 - MDRD (N=169, 132) | 45.2 (15.3) | 48.0 (13.5)
  Week 1 - CG (N=224, 165) | 35.0 (13.9) | 39.6 (15.7)
  Week 14 - CG (N=181, 143) | 35.9 (15.2) | 41.6 (16.9)
  Week 26 - CG (N=167, 132) | 37.4 (15.6) | 41.8 (16.8)

5. Secondary Outcome: Physical Performance: Speed Walked or Wheeled in a Maximum of 10 Minutes at Each Visit
Description: Physical performance was measured for all patients with CKD (defined as estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73m^2). The average speed a participant walked, with or without an assistive device, and stand-by assistance of one person or propelled themselves in their wheelchair with or without the use of their feet, over level ground, up to 10 minutes with up to two 30 second rest periods.
Time Frame: Weeks 2, 14 and 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Mean (Standard Deviation); unit: feet per minute
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 208 | 152
feet per minute
  Week 2 (N=208, 152) | 51.2 (40.4) | 61.9 (51.4)
  Week 14 (N=172, 132) | 51.0 (41.6) | 70.1 (59.0)
  Week 26 (N=158, 123) | 49.9 (42.2) | 66.5 (62.3)

6. Secondary Outcome: Physical Performance: Duration Walked or Wheeled at Each Visit
Description: The duration a participant was able to walk or propel themselves in a wheelchair during 10 minutes.
Time Frame: Weeks 2, 14, 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 208 | 152
minutes
  Week 2 (N=208, 152) | 6.4 (3.3) | 6.2 (3.1)
  Week 14 (N=173, 133) | 6.5 (3.1) | 6.4 (3.2)
  Week 26 (N=158, 124) | 6.6 (3.1) | 6.0 (3.2)

7. Secondary Outcome: Physical Performance: Time to Rise From Sitting to Standing
Description: Participants were asked to stand from a seated position so that knees approximated full extension. Timing began from the point that the participant initiated the standing behavior to the point he/she was on his/her feet with knees at approximately full extension.
Time Frame: Weeks 2, 14, 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 171 | 133
seconds
  Week 2 (N=171, 133) | 3.0 [2.0 to 6.0] | 3.0 [2.0 to 6.0]
  Week 14 (N=134, 114) | 2.5 [1.5 to 5.8] | 3.0 [1.7 to 5.0]
  Week 26 (N=125, 108) | 3.0 [1.2 to 6.0] | 3.0 [1.5 to 4.6]

8. Secondary Outcome: Physical Performance: Grip Strength
Description: Grip strength was measured using an adjustable, hand-held, hydraulic grip strength dynamometer. While seated, participants were asked to grip the 2 bars of the dynamometer in their hand and slowly squeeze as hard as they can; then relax. The highest of three measurements was recorded.
Time Frame: Weeks 2, 14, 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Mean (Standard Deviation); unit: pound-force
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 215 | 154
pound-force
  Week 2 (N=215, 154) | 29.6 (17.4) | 31.8 (16.9)
  Week 14 (N=182, 140) | 29.8 (17.3) | 32.5 (17.1)
  Week 26 (N=166, 129) | 29.0 (16.9) | 29.8 (17.4)

9. Secondary Outcome: Physical Performance: Lower Extremity Strength, Left Leg.
Description: Lower extremity strength test measures the maximum amount of weight a participant can lift one time throughout his/her range of motion. While supine, and using adjustable cuff weights, participants were asked to bend at their hip and knee and draw their heel along the bed towards their buttocks.
Time Frame: Weeks 2, 14, 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 211 | 151
pounds
  Week 2 (N=211, 151) | 5.3 (4.1) | 6.1 (4.1)
  Week 14 (N=174, 136) | 5.3 (4.4) | 6.6 (4.6)
  Week 26 (N=159, 125) | 5.6 (4.5) | 6.4 (4.5)

10. Secondary Outcome: Physical Performance: Lower Extremity Strength, Right Leg
Description: as for outcome 9
Time Frame: Weeks 2, 14, 26
Population: Enrolled patients with CKD and non-missing data at each time point (indicated by "N").
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | CKD With Anemia | CKD With no Anemia
Number analyzed (Participants) | 212 | 151
pounds
  Week 2 (N= 212, 151) | 5.3 (4.0) | 6.3 (4.0)
  Week 14 (N=174, 136) | 5.2 (4.0) | 6.1 (4.1)
  Week 26 (N=159, 125) | 5.6 (4.5) | 6.5 (4.5)

ADVERSE EVENTS:
Description: Adverse Events were not collected for this observational protocol.
Arm/Group | No CKD or Anemia | CKD With Anemia | CKD With no Anemia | No CKD, But Anemia
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
21 subjects could not be classified into the defined groups because of missing lab values at enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.